CLINICAL TRIAL: NCT03682926
Title: EFFECT OF A PROTOCOL Electrostimulation for Urinary Incontinence and Its Influence on WOMEN 'S QUALITY OF LIFE
Brief Title: Electrostimulation PROTOCOL Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, ROSANA CRISTINA PEREIRA DE ANDRADE, Dra, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROAND2015
Record Dates: First submitted 2015-03-11; First posted 2018-09-25 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Female Stress Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- electrostimulation individualized (Experimental): Selective electrostimulation for tonic fiber, phasic fiber FIa and FIIb and different stimulus times. Muscle fibers (Tonic) with a frequency of 20Hz, pulse width (t) of 700μs to 1ms, time of rise and fall of the wave of 1.0 seconds, duration of contraction and repetition was based on the perineal evaluation But the resting time was twice as long as sustained. For the IIa (phasic) fibers the frequency was 50 Hz with a pulse width of 400μs to 500μs, for 3 seconds of sustentation and 6 seconds of relaxation, time of rise of 0,5 seconds and 0,5 seconds of descent. E for type IIb (phasic) fibers, 80 Hz frequency, pulse width 250μs to 400μs, 1 second contraction for 3 seconds rest and 0.2 seconds rise and fall time.
  Interventions: Other: Electro-stimulation
- electrostimulation with fixed protocol (Active Comparator): Intervention -Electro-stimulate all fibers with a single electrical parameter. Pulse width 700μs, rise and fall time of 2 seconds each, sustain time of 4 seconds and rest 8 seconds for 20 minutes, the intensity will be modulated, as in the previous group by patient tolerance in milliamperes.
  Interventions: Other: Electro-stimulation

INTERVENTIONS:
Other: Electro-stimulation — Intracavitary electrostimulation with Quark medical vaginal electrode for perineal muscle strengthening protocol.
  Other Names: electro physical therapy; dualpex 961 quark

SUMMARY:
To verify the effect of an adapted electrostimulation (EE) protocol for stress and mixed urinary incontinence (SUI / M) and its impact on quality of life (QoL)

DETAILED DESCRIPTION:
Controlled and randomized clinical trial performed at the Physiotherapy Outpatient Clinic at the Magalhães Neto Pavilion of ComHUPES / UFBA. Women aged between 30 and 65 years and diagnosis of SUI / IUM. The patients were allocated to two groups (GA) submitted to selective electrostimulation for tonic fiber, phasic fibers IIa / IIb and different times of electrical stimulation; (GB) used 50hz for all fibers by 20mm, both answered the questionnaire King's Health Questionnaire (KHQ).

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 30 and 65
* With diagnosis of stress urinary incontinence and / or mixed
* Perineal muscle weakness
* Accepted to sign the TCLE

Exclusion Criteria:

* Women with neurological changes
* Pregnant women
* IUD use
* Pacemaker
* Genitourinary tract infection
* Cancer
* Refuse to sign the TCLE

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
contractile function of the perineal musculature | 3 months
  Perineal muscle function evaluated subjectively by vaginal touch using the PERFECT system to measure strength (graded from 0 to 5), strength (holding capacity of contraction recorded in seconds) and number of contractions of tonic and phasic fibers (ability to repeat muscle contractions perineal). Objectively, the vaginal cones were used to determine which load the patient was able to support (kit with 5 cones with weights ranging from 20 to 70g)

SECONDARY OUTCOMES:
King's Health Questionnaire | 3 months
  It allows qualitative evaluation of the impact of urinary incontinence on the quality of life of women, it is responsible for 20 questions, divided into 8 domains, in addition to these domains, there are two other independent scales: the first evaluates the severity of UI (severity measures) and the second, the presence and intensity of urinary symptoms through the scale of urinary symptoms (VAS) where there is a graduation from 0 to 10, where the higher the score, the higher the severity

IPD SHARING:
Plan to Share IPD: No